CLINICAL TRIAL: NCT00373529
Title: A Phase II Study of Single Agent Clofarabine in Previously Untreated Older Adult Patients With Acute Myelogenous Leukemia (AML) for Whom Standard Induction Chemotherapy is Unlikely to be of Benefit
Brief Title: A Study of Clofarabine for Older Patients With Newly Diagnosed Acute Myelogenous Leukemia (AML) (CLASSIC II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO24300606
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Acute Myelogenous Leukemia; Acute Myeloid Leukemia
Keywords: Acute myelogenous leukemia; Acute myeloid leukemia; newly Diagnosed AML; Clofarabine; CLASSIC II; CLO243
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine (Experimental): Participants received an induction cycle of clofarabine 30 mg/m^2/day intravenous infusion for 5 consecutive days. Participants could then receive up to 5 additional cycles, repeated minimally every 28 days, of clofarabine 20 mg/m^2/day intravenous infusion for 5 consecutive days.
  Interventions: Drug: clofarabine

INTERVENTIONS:
Drug: clofarabine — Induction cycle 1: cycle 1 of clofarabine 30 mg/m^2/day as a 1-hour intravenous infusion for 5 consecutive days.
  Reinduction (cycle 2) and/or Consolidation cycles (cycles 2-6): cycles repeated minimally every 28 days, of clofarabine 20 mg/m^2/day as a 1-hour intravenous infusion for 5 consecutive days.
  Other Names: clolar

SUMMARY:
Clolar (clofarabine injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed acute lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens.

This study will evaluate the efficacy of clofarabine in elderly patients with acute myelogenous leukemia (AML) who are unlikely to benefit from treatment with intensive chemotherapy regimens (cytarabine and anthracycline based regimens) used in younger patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML (de novo, secondary or with an antecedent hematologic disorder [AHD])
* Age ≥ 60 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Presence of at least one adverse prognostic factor: Age ≥ 70 years; or AHD; or ECOG performance status of 2; or Intermediate or unfavorable (i.e., adverse) karyotype defined as any cytogenetic profile except the presence of any of the following:

  * t(8;21)(q22;q22)
  * inv(16)(p13;q22 or t(16;16)(p13;q22)
  * t(15;17)(q22;q12) and variants.
* Adequate renal and hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN; and Serum creatinine ≤ 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease (MDRD) equation
* Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 40% or left ventricular fractional shortening ≥ 22%

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Prior treatment with clofarabine
* Prior treatment for AML or an antecedent hematologic disorder
* Prior hematopoietic stem cell transplant (HSCT)
* Prior radiation therapy to the pelvis
* Investigational agent received within 30 days prior to the first dose of study drug
* Ongoing uncontrolled systemic infection
* Diagnosis of another malignancy, unless the patient has been disease-free for at least 5 years following the completion of curative intent therapy with the following exceptions: Patients with treated non-melanoma skin cancer, in-situ carcinoma or cervical intraepithelial neoplasia regardless of disease-free duration are eligible for this study if definitive treatment for the condition has been completed; Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on PSA value are eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* Clinical evidence of central nervous system (CNS) involvement
* Severe concurrent medical condition or psychiatric disorder that would preclude study participation
* Positive human immunodeficiency virus (HIV) test

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (20):
- United States (20):
  - Mayo Clinical Hospital, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Scripps Cancer Center, San Diego, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of MD Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University - HSC, Morgantown, West Virginia

REFERENCES:
- [Result] Kantarjian HM, Erba HP, Claxton D, Arellano M, Lyons RM, Kovascovics T, Gabrilove J, Craig M, Douer D, Maris M, Petersdorf S, Shami PJ, Yeager AM, Eckert S, Abichandani R, Faderl S. Phase II study of clofarabine monotherapy in previously untreated older adults with acute myeloid leukemia and unfavorable prognostic factors. J Clin Oncol. 2010 Feb 1;28(4):549-55. doi: 10.1200/JCO.2009.23.3130. Epub 2009 Dec 21. PMID 20026805

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 129 patients were screened and 116 participants enrolled/treated at 20 sites.
Period: Overall Study
Arm/Group | Clofarabine
Started | 116
Full Analysis Set | 112 (3 Failed Independent Confirmation of AML; 1 consent violation)
Completed | 8 (Completed: initiated full 6 cycles of treatment. Not Completed: initiated <6 cycles of treatment)
Not Completed | 108
Not completed — Physician Decision | 19
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 7
Not completed — Treatment failure | 36
Not completed — Disease recurrence | 10
Not completed — Death | 16
Not completed — Need for treatment prohibited by study | 1
Not completed — Other | 8
Not completed — Failed independent confirmation of AML | 3
Not completed — Consent violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (5.92)
Age, Continuous [Median (Full Range); unit: years] | 71.0 [60 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 52
Race [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 98
  Other | 2
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 108
Height [Mean (Standard Deviation); unit: cm] | 166.50 (10.366)
Weight [Mean (Standard Deviation); unit: kg] | 78.45 (18.191)
Age at Enrollment [Number; unit: participants] — Being 70 years old or older is considered an adverse prognostic factor.
  participants
    >= 70 years | 69
    < 70 years | 43
Antecedent Hematologic Disorder [Number; unit: participants] — The most common risk factor for acute myelogenous leukemia (AML) is the presence of an antecedent hematologic disorder.
  participants
    Yes | 41
    No | 67
    Not reported | 4
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Another prognostic factor. Eastern Cooperative Oncology Group Performance Status (ECOG PS) is a scale ranging from 0-5, with 0=fully active, 1=capable of light work, 2=no work but all self-care, 3=limited self-care, 4=completely disabled, 5=dead.
  participants
    ECOG 5 | 0
    ECOG 4 | 0
    ECOG 3 | 0
    ECOG 2 | 25
    ECOG 1 | 66
    ECOG 0 | 21
Karyotype [Number; unit: participants] — A favorable cytogenetic karyotype is associated with a positive prognostic outcome; an unfavorable cytogenetic karyotype is associated with a negative prognostic outcome. An intermediate karyotype is typically associated with a better outcome than a favorable karyotype, but also associated with a worse outcome compared to a favorable karyotype.
  participants
    Intermediate | 46
    Unfavorable | 62
    Favorable | 0
    Not reported | 4
Participants Summarized by Number of Adverse Prognostic Factors [Number; unit: participants] — Participant counts by the number of adverse prognostic factors, which include age >= 70 years, antecedent hematologic disorder = Yes, ECOG = 2, and karyotype = intermediate or unfavorable.
  participants
    0 Adverse Prognostic Factors | 0
    1 Adverse Prognostic Factor | 25
    2 Adverse Prognostic Factors | 45
    3 Adverse Prognostic Factors | 40
    4 Adverse Prognostic Factors | 2
Participants Summarized by Number of Adverse Prognostic Factors Excluding Intermediate Karyotype [Number; unit: participants] — Participant counts by the number of adverse prognostic factors, which include age >= 70 years, antecedent hematologic disorder = Yes, ECOG = 2, and karyotype = unfavorable.
  participants
    0 Adverse Prognostic Factors | 7
    1 Adverse Prognostic Factor | 42
    2 Adverse Prognostic Factors | 35
    3 Adverse Prognostic Factors | 27
    4 Adverse Prognostic Factors | 1
Secondary acute myeloid leukemia (AML) at baseline [Number; unit: participants] — The diagnosis of secondary AML is based upon investigator judgment regarding prior ionizing radiation and/or chemotherapy.
  participants
    Yes | 11
    No | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Overall Remission (OR) After No More Than Two Cycles (Approximately Month 2)
Description: Best response was assessed by the Independent Response Review Panel(IRRP) after two cycles of treatment. Overall remission(OR) is the sum of complete remission(CR) and complete remission in the absence of platelet recovery(CRp). CR includes normal values for peripheral blood cell counts (absolute neutrophil and platelet) and leukemic blast cells from bone marrow biopsy or aspirate, and absence of extramedullary disease. Partial remission(PR) includes recovery of peripheral blood cells with improved but still abnormal values in leukemic blast cells.
Time Frame: approximately Month 2
Population: Full analysis set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 112
percentage of participants
  Overall Remission (OR=CR+CRp) | 45.5
  Complete Remission (CR) | 37.5
  Complete Remission w/o platelet recovery (CRp) | 8.0
  Partial Remission (PR) | 3.6
  Treatment Failure (TF) | 50.9

2. Secondary Outcome: Kaplan Meier Estimate for Duration of Remission (DOR)
Description: DOR was defined as the number of days from achievement of OR as assessed by the Independent Response Review Panel (IRRP) until IRRP-determined disease recurrence or death (any cause), plus 1 day. Participants who initiated alternative antileukemic treatment while in remission were censored on the date the therapy was initiated or on the date of last follow-up.
Time Frame: Up to 2 years
Population: Full analysis set (FAS) of participants who achieved remission.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Clofarabine
Number analyzed (Participants) | 51
weeks | 55.6 [33.1 to 82.9]

3. Secondary Outcome: Kaplan Meier Estimate for Disease-free Survival (DFS)
Description: DFS was defined as the number of days from achievement of IRRP-determined overall response until IRRP-determined disease recurrence or death (any cause), regardless of intervening alternative antileukemic treatment, plus 1 day.
Time Frame: Up to 2 years
Population: Full analysis set (FAS) of participants who achieved remission.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Clofarabine
Number analyzed (Participants) | 51
weeks | 43.8 [27.6 to 60.7]

4. Secondary Outcome: Kaplan Meier Estimates for Overall Survival (OS)
Description: OS was defined as the number of days from first dose of clofarabine until death for all participants, plus 1 day.
Time Frame: Up to 2 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Clofarabine
Number analyzed (Participants) | 112
weeks | 40.7 [28.3 to 52.0]

5. Secondary Outcome: Overall Participant Counts Summarizing Adverse Events (AEs) During the Treatment and Follow-up Periods
Description: Participants with AEs that occurred during the treatment and follow-up periods. AEs were classified according to severity (graded using National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 3.0) and relationship to study drug. Treatment emergent is defined as any event that either first presents after baseline or worsens in severity after baseline.
  NCI Common Terminology Criteria for Severity:
  Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5= Death related to AE
Time Frame: Up to 2 years
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 112
participants
  Treatment-emergent AEs (TEAE) | 112
  Treatment-emergent AEs related to study drug | 108
  Treatment-emergent serious AEs | 76
  Treatment-emergent serious AEs related to drug | 41
  Discontinued due to AEs | 7
  Died w/i treatment period-w/i 45 days of last dose | 22
  Died due to drug-related AEs | 4
  Died within 30 days of first dose | 11
  Died w/i 30 days of first dose due to related AEs | 3
  Grade 1: maximum severity rating for any TEAE | 2
  Grade 2: maximum severity rating for any TEAE | 6
  Grade 3: maximum severity rating for any TEAE | 46
  Grade 4: maximum severity rating for any TEAE | 34
  Grade 5: maximum severity rating for any TEAE | 24

6. Secondary Outcome: Percentage of Participants Who Died Within Thirty Days of Treatment (30-day Mortality Rate)
Description: Percentage of participants who died within 30 days of the first dose of study drug, regardless of cause.
Time Frame: up to Day 30
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 112
percentage of participants | 9.8

7. Other Pre Specified Outcome: Number of Participants Achieving Overall Remission After A Maximum of Two Cycles by Subgroup of Baseline Prognostic Factors
Description: The number of participants within each subgroup of baseline prognostic factors of the full analysis set who achieved a best response of either a complete response (CR) or a complete response in the absence of platelet recovery (CRp) as determined by the Independent Response Review Panel following a maximum of two cycles of treatment.
Time Frame: approximately Month 2
Population: Full analysis set (FAS) of participants who achieved remission and had baseline prognostic factor
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 112
participants
  Age >=70 (n=69) | 27
  Age <70 (n=43) | 24
  Antecedent hematologic disorder - Yes (n=41) | 21
  Antecedent hematologic disorder - No (n=67) | 29
  Antecedent hematologic disorder-Not reported (n=4) | 1
  ECOG Performance Status = 0-1 (n=87) | 43
  ECOG Performance Status = 2 (n=25) | 8
  Karyotype = Intermediate (n=46) | 25
  Karyotype = Unfavorable (n=62) | 26
  Karyotype = Not Reported (n=4) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Clofarabine
Serious Adverse Events (participants affected / at risk) | 76/112
Other Adverse Events (participants affected / at risk) | 112/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (N=112)
Anaemia (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 28
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 7
Cardiac failure congestive (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Haematemesis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Fatigue (General disorders) | 2
Multi-organ failure (General disorders) | 2
Organ failure (General disorders) | 1
Pyrexia (General disorders) | 1
Abscess intestinal (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 4
Bacterial infection (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 4
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 4
Clostridial infection (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 6
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Enterococcal bacteraemia (Infections and infestations) | 3
Enterococcal sepsis (Infections and infestations) | 2
Escherichia bacteraemia (Infections and infestations) | 1
Herpes oesophagitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 2
Oral bacterial infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 16
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia chlamydial (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 3
Pseudomonal sepsis (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Respiratory moniliasis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 6
Septic shock (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Sinusitis bacterial (Infections and infestations) | 1
Sinusitis fungal (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 3
Staphylococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Urinary tract infection bacterial (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Bacterial test (Investigations) | 1
Bacterial test positive (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Staphylococcus test positive (Investigations) | 1
Troponin I increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Fluid overload (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Cerebrovascular accident (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 9
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2
Jugular vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clofarabine (N=112)
Anaemia (Blood and lymphatic system disorders) | 12
Coagulopathy (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 50
Hypergammaglobulinaemia (Blood and lymphatic system disorders) | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Lymph node calcification (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 5
Lymphocytic infiltration (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 21
Pancytopenia (Blood and lymphatic system disorders) | 4
Platelet disorder (Blood and lymphatic system disorders) | 1
Splenic granuloma (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 18
White blood cell disorder (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 4
Aortic valve disease (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 11
Bradycardia (Cardiac disorders) | 4
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardiomegaly (Cardiac disorders) | 8
Cardiomyopathy (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 1
Diastolic dysfunction (Cardiac disorders) | 2
Dilatation atrial (Cardiac disorders) | 1
Dilatation ventricular (Cardiac disorders) | 2
Electromechanical dissociation (Cardiac disorders) | 1
Extrasystoles (Cardiac disorders) | 2
Heart valve incompetence (Cardiac disorders) | 1
Left atrial dilatation (Cardiac disorders) | 5
Left ventricular hypertrophy (Cardiac disorders) | 4
Mitral valve calcification (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 6
Pericardial cyst (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 11
Pulmonary valve incompetence (Cardiac disorders) | 2
Right atrial dilatation (Cardiac disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 7
Supraventricular extrasystoles (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 25
Tricuspid valve incompetence (Cardiac disorders) | 3
Ventricular extrasystoles (Cardiac disorders) | 3
Ventricular hypokinesia (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Ear congestion (Ear and labyrinth disorders) | 2
Ear discomfort (Ear and labyrinth disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Hypoacusis (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 5
Adrenal insufficiency (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secre (Endocrine disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 3
Conjunctival hyperaemia (Eye disorders) | 1
Conjunctival oedema (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 3
Diplopia (Eye disorders) | 2
Dry eye (Eye disorders) | 8
Eye disorder (Eye disorders) | 1
Eye oedema (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid disorder (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Mydriasis (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Photophobia (Eye disorders) | 2
Pinguecula (Eye disorders) | 1
Scleral oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 6
Visual acuity reduced (Eye disorders) | 1
Visual impairment (Eye disorders) | 4
Vitreous haemorrhage (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 27
Abdominal pain lower (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 6
Abdominal tenderness (Gastrointestinal disorders) | 8
Anal fissure (Gastrointestinal disorders) | 1
Anal pruritus (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1
Caecitis (Gastrointestinal disorders) | 1
Chapped lips (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 48
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 72
Diverticulum (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 16
Dysphagia (Gastrointestinal disorders) | 10
Epigastric discomfort (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 5
Faecaloma (Gastrointestinal disorders) | 1
Faeces hard (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 8
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Gingival bleeding (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 4
Glossodynia (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 4
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 15
Hiatus hernia (Gastrointestinal disorders) | 5
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 4
Lip blister (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 6
Lip swelling (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 2
Loose tooth (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 3
Mouth haemorrhage (Gastrointestinal disorders) | 10
Mouth ulceration (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 85
Odynophagia (Gastrointestinal disorders) | 3
Oesophagitis (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 5
Pancreatic atrophy (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 5
Proctalgia (Gastrointestinal disorders) | 1
Proctitis ulcerative (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Rectal prolapse (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 2
Saliva altered (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 12
Tongue discolouration (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Tongue haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 63
Asthenia (General disorders) | 22
Catheter site discharge (General disorders) | 4
Catheter site erythema (General disorders) | 21
Catheter site haematoma (General disorders) | 4
Catheter site haemorrhage (General disorders) | 5
Catheter site inflammation (General disorders) | 2
Catheter site oedema (General disorders) | 1
Catheter site pain (General disorders) | 13
Catheter site rash (General disorders) | 2
Catheter site related reaction (General disorders) | 2
Chest discomfort (General disorders) | 5
Chest pain (General disorders) | 5
Chills (General disorders) | 40
Device occlusion (General disorders) | 2
Discomfort (General disorders) | 1
Face oedema (General disorders) | 1
Facial pain (General disorders) | 2
Fatigue (General disorders) | 40
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 1
Generalised oedema (General disorders) | 5
Granuloma (General disorders) | 1
Hypothermia (General disorders) | 1
Infusion site induration (General disorders) | 1
Infusion site urticaria (General disorders) | 1
Injection site haematoma (General disorders) | 1
Irritability (General disorders) | 2
Local swelling (General disorders) | 1
Localised oedema (General disorders) | 3
Malaise (General disorders) | 9
Mucosal dryness (General disorders) | 3
Mucosal inflammation (General disorders) | 18
Non-cardiac chest pain (General disorders) | 4
Oedema (General disorders) | 8
Oedema peripheral (General disorders) | 63
Pain (General disorders) | 12
Pyrexia (General disorders) | 44
Swelling (General disorders) | 1
Temperature intolerance (General disorders) | 1
Thrombosis in device (General disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 4
Gallbladder disorder (Hepatobiliary disorders) | 2
Gallbladder oedema (Hepatobiliary disorders) | 2
Granulomatous liver disease (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 3
Hepatic lesion (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 10
Jaundice (Hepatobiliary disorders) | 2
Portal hypertension (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 6
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Alpha haemolytic streptococcal infection (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 4
Bacterial infection (Infections and infestations) | 3
Bacteroides infection (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 6
Chronic sinusitis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 4
Clostridium difficile colitis (Infections and infestations) | 7
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 4
Device related sepsis (Infections and infestations) | 1
Enterobacter infection (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 3
Enterococcal infection (Infections and infestations) | 5
Escherichia bacteraemia (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal candidiasis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 3
Hepatitis b (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Jc virus infection (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Morganella infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Neutropenic infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 18
Oral herpes (Infections and infestations) | 5
Oral viral infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 17
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 3
Post procedural cellulitis (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Respiratory moniliasis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Sinusitis fungal (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 8
Staphylococcal infection (Infections and infestations) | 4
Streptococcal bacteraemia (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 5
Urinary tract infection bacterial (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 17
Excoriation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 3
Muscle strain (Injury, poisoning and procedural complications) | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 3
Pocket erosion (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 7
Renal haematoma (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 5
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 26
Antibiotic resistant staphylococcus test (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 24
Bacterial test positive (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 5
Blood amylase increased (Investigations) | 5
Blood bicarbonate decreased (Investigations) | 1
Blood bicarbonate increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 7
Blood chloride decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 13
Blood culture positive (Investigations) | 2
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 3
Blood phosphorus decreased (Investigations) | 2
Blood phosphorus increased (Investigations) | 2
Blood potassium decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood urine present (Investigations) | 1
Bone density increased (Investigations) | 1
Brain natriuretic peptide increased (Investigations) | 3
Breath sounds abnormal (Investigations) | 10
Cardiac murmur (Investigations) | 10
Chest x-ray abnormal (Investigations) | 3
Clostridium test positive (Investigations) | 1
Coagulation time prolonged (Investigations) | 1
Culture urine positive (Investigations) | 2
Electrocardiogram qt prolonged (Investigations) | 3
Electrocardiogram st segment abnormal (Investigations) | 1
Electrocardiogram st segment depression (Investigations) | 1
Electrocardiogram t wave abnormal (Investigations) | 4
Enterococcus test positive (Investigations) | 3
Eosinophil count increased (Investigations) | 1
Face and mouth x-ray abnormal (Investigations) | 1
Fungal test positive (Investigations) | 1
Haemoglobin (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate irregular (Investigations) | 4
Heart sounds abnormal (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Lipase increased (Investigations) | 7
Liver function test abnormal (Investigations) | 3
Liver palpable subcostal (Investigations) | 1
Occult blood positive (Investigations) | 3
Oxygen saturation decreased (Investigations) | 1
Protein total decreased (Investigations) | 1
Pulmonary arterial pressure increased (Investigations) | 1
Right ventricular systolic pressure incr (Investigations) | 1
Streptococcus test positive (Investigations) | 2
Transaminases increased (Investigations) | 8
Troponin I (Investigations) | 1
Troponin I increased (Investigations) | 1
Urine analysis abnormal (Investigations) | 1
Urine output decreased (Investigations) | 2
Weight decreased (Investigations) | 17
Weight increased (Investigations) | 3
White blood cell count decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 45
Dehydration (Metabolism and nutrition disorders) | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Fluid imbalance (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 18
Fluid retention (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 36
Hypomagnesaemia (Metabolism and nutrition disorders) | 14
Hyponatraemia (Metabolism and nutrition disorders) | 9
Hypophagia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 13
Increased appetite (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1
Podagra (Metabolism and nutrition disorders) | 1
Polydipsia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 6
Vitamin k deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Back pain (Musculoskeletal and connective tissue disorders) | 25
Bone lesion (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 13
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 11
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemic retinopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Spinal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 26
Dizziness postural (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 8
Embolic stroke (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Facial palsy (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 45
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 6
Orthostatic intolerance (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 11
Parosmia (Nervous system disorders) | 2
Peroneal nerve palsy (Nervous system disorders) | 1
Poor quality sleep (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 2
Radial nerve palsy (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 10
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 6
Tension headache (Nervous system disorders) | 1
Tongue paralysis (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 5
Abnormal behaviour (Psychiatric disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 26
Claustrophobia (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 25
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 14
Disorientation (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 4
Hallucination, visual (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 46
Mental status changes (Psychiatric disorders) | 8
Mood altered (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 2
Panic attack (Psychiatric disorders) | 1
Phonophobia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
Bladder dilatation (Renal and urinary disorders) | 3
Bladder hypertrophy (Renal and urinary disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Bladder spasm (Renal and urinary disorders) | 3
Chromaturia (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 6
Haematuria (Renal and urinary disorders) | 9
Hydronephrosis (Renal and urinary disorders) | 1
Ketonuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 4
Oliguria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 4
Polyuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 8
Renal failure acute (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 11
Urinary retention (Renal and urinary disorders) | 5
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Oedema genital (Reproductive system and breast disorders) | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Penile swelling (Reproductive system and breast disorders) | 2
Prostatomegaly (Reproductive system and breast disorders) | 1
Scrotal haematocoele (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 3
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 34
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1
Egobronchophony (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 5
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 14
Rales (Respiratory, thoracic and mediastinal disorders) | 19
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 9
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 3
Blood blister (Skin and subcutaneous tissue disorders) | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 9
Ecchymosis (Skin and subcutaneous tissue disorders) | 19
Erythema (Skin and subcutaneous tissue disorders) | 14
Exfoliative rash (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2
Leukoplakia (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 7
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndr (Skin and subcutaneous tissue disorders) | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 29
Pruritus (Skin and subcutaneous tissue disorders) | 26
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 52
Rash erythematous (Skin and subcutaneous tissue disorders) | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 15
Rash macular (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Rash papular (Skin and subcutaneous tissue disorders) | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 6
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 6
Skin mass (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 2
Skin oedema (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 5
Fasciotomy (Surgical and medical procedures) | 1
Leg amputation (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 3
Aortic calcification (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 2
Capillary leak syndrome (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Flushing (Vascular disorders) | 13
Haematoma (Vascular disorders) | 8
Haemorrhage (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 22
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 32
Orthostatic hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 6
Pallor (Vascular disorders) | 4
Peripheral coldness (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.